CLINICAL TRIAL: NCT05172817
Title: A Prospective, Randomized, Double Blind, Active Controlled Study to Compare PK & Safety of Biosimilar Adalimumab (Advixa) 40 mg/ 0.4 ml of Incepta Pharmaceuticals Ltd. With Humira 40 mg/ 0.4ml of Abbvie Ltd. in Healthy, Adult, Human Subject by Single Subcutaneous Injection Followed by Efficacy & Safety Study in Patients With Rheumatoid Arthritis
Brief Title: Study to Compare PK & Safety of Advixa With Humira in Healthy, Adult Subject Followed by Efficacy & Safety Study in RA Patients
Acronym: ACT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute for Developing Science and Health Initiatives, Bangladesh (Other)
Collaborators: Universal Medical College Hospital, Bangladesh (Unknown); Green Life Center for Rheumatic Care & Research, Bangladesh (Unknown); Incepta Pharmaceuticals Ltd, Bangladesh (Unknown)
Responsible Party: Principal Investigator, Dr. Mohammad Badrul Anam, Principal Investigator, Institute for Developing Science and Health Initiatives, Bangladesh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDE-21-005
Record Dates: First submitted 2021-09-28; First posted 2021-12-29 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Pharmacokinetics; Safety; Efficacy; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advixa (Experimental): Generic name: Adalimumab Dosage form: Injectable Route of Administration: Subcutaneous Dosage: 40mg/0.4mL Frequency: Once in 2 weeks Duration: Single dose for Phase 2 and 3 months for Phase 3
  Interventions: Drug: Advixa (Adalimumab)
- Humira (Active Comparator): Generic name: Adalimumab Dosage form: Injectable Route of Administration: Subcutaneous Dosage: 40mg/0.4mL Frequency: Once in 2 weeks Duration: Single dose for Phase 2 and 3 months for Phase 3
  Interventions: Drug: Advixa (Adalimumab)

INTERVENTIONS:
Drug: Advixa (Adalimumab) — Injection Advixa(Adalimumab) 40 mg/ 0.4 ml will be administered subcutaneously to the participants by trained medical personnel. Single dose for phase 2 and biweekly for 3 months for phase 3.

SUMMARY:
Adalimumab is a recombinant monoclonal antibody (IgG1 subclass) against human TNF-α (Tumor Necrosis Factor-alpha). It is an immunosuppressive medication predominantly used to treat rheumatoid arthritis autoimmune disease. It is also used for the treatment of psoriatic arthritis, ankylosing spondylitis, and Crohn's disease etc. Adalimumab binds specifically to TNF-α and blocks its general cytokine effects, thereby reducing TNF-induced inflammation and halting tissue destruction. Adalimumab was approved for medical use in the United States in 2002. It is on the World Health Organization's List of Essential Medicines. It is available as a biosimilar medication. In 2017, it was the 169th most commonly prescribed medication in the United States, with more than three million prescriptions. Adalimumab is an expensive product which is indicated in rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, Crohn's disease, etc. Each patient will be provided the study drug free of cost in this study which will benefit them immensely.

The advent of therapeutic monoclonal antibodies has given a major boost to the treatment of individuals suffering from autoimmune disorders, including rheumatoid arthritis. Adalimumab is one such therapeutic monoclonal antibody used for treatment of rheumatoid arthritis marketed with brand name Humira by Abbvie Ltd. (USA) was the only adalimumab biosimilar available for patients in Bangladesh until recently. Incepta Pharmaceuticals Ltd. Bangladesh has introduced Bangladesh's first locally manufactured adalimumab biosimilar Advixa that is available at a fraction of Humira's cost. This study aims to evaluate the pharmacokinetics, safety and efficacy of the Adalimumab biosimilar (Advixa) in comparison to Adalimumab (Humira) as reference. The biosimilar Advixa being a local product will a cost-effective alternative to imported drugs currently available in the market.

Objectives of the Protocol

General objectives-

1. To assess the Pharmacokinetic between Test Product (A): Adalimumab (Advixa) 40 mg/ 0.4 ml of Incepta Pharmaceuticals Ltd of Bangladesh and the corresponding Reference Product

   (B): Humira 40 mg/ 0.4ml of Abbvie Ltd in normal, healthy, adult, human subjects in a Parallel group study.
2. To evaluate the safety between two products.
3. To assess efficacy, tolerability and safety of biosimilar adalimumab (Advixa, Incepta) in compared with reference adalimumab (Humira, AbbVie) in patients with moderate to severe rheumatoid arthritis (RA).

Specific objectives-

1. Pharmacokinetic (PK) Parameters: For Cmax and AUC0-t the 90% confidence interval for the ratio of the test and reference products should be contained within the acceptance interval of 80.00-125.00%.
2. Safety assessment: Evaluation and comparison between references vs. test drug in terms of safety end point.
3. Efficacy assessment: The primary endpoints will be -

   1. Proportion of patients with an ACR20 response in both the treatment groups at week 12.
   2. Evaluation and comparison of safety between references vs. test drug.

The secondary endpoints will be -

1. Change in Disease Activity Score of 28 joints - CRP (DAS28-CRP),
2. Proportion of patient with an ACR50 response and
3. Proportion of patients with an ACR70 response in both the treatment groups at week 12.

DETAILED DESCRIPTION:
This study will have two parts, Part A and Part B. Part A will be conducted in apparently healthy, adult human subjects to evaluate the safety between test and reference products and to assess the Pharmacokinetic (PK) parameters. After the Part A completed the result will be reviewed by DSMB. Then only after successful DSMB favorable opinion the Part B of the study will start. Part B will be conducted in patients with moderate to severe rheumatoid arthritis (RA) to assess efficacy, tolerability and safety between test and reference products.

Descriptions for Part A and Part B of the study are as follows-

PART A

A Prospective, Randomized, Double blind, Parallel-group, Active controlled, Pk and safety study in Healthy, Adult, Human Subject by single subcutaneous injection. The sample size is 40. Single subcutaneous injection of 40 mg/ 0.4 ml dose of test or reference product will be administered as per the randomization schedule. In patient facility will be at least 12 hours prior to drug administration until 48 hrs post dose. The duration of the study will be 3 months. Housing 2 days, active / solicited safety follow-up for Adverse Events (either home visit or telephone call) will be performed from day 3 to day 8 and passive / un-solicited safety follow-up (spontaneous AE reporting by subject) will be performed for day 9 to day 64. Clinic visit at day 64 and day 90 for Safety evaluation.

Subjects will be screened for the inclusion/exclusion criteria based on: Demographic data, BMI, clinical history, physical examination (including vital signs), Haemogram, Random blood sugar, Serum bilirubin Total/Direct/Indirect, BUN, Serum urea, ALT (SGPT) blood, AST (SGOT) blood, Alkaline phosphatase serum, Serum creatinine, ECG, BNP, Chest X-ray (P/A view) (if required based on any significant past medical history and/or positive finding in respiratory system examination), Quantiferon TB gold plus, serology (HIV, hepatitis B and hepatitis C), Urinalysis, Amphetamines urine, Benzodiazepines urine, COVID-19 qRT-PCR. Breath alcohol test will be done during the screening.

For female volunteers: In addition to the above tests, urine pregnancy test will be done at the time of screening.

Any other test(s) if required will be done as per the suggestion given by the principal investigator or co-investigator.

Blood samples will be collected for serum drug concentration measurements at Time points: Pre-dose (-15 min) and post-dose 04, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 360, 528, 696, 864, 1032, 1200, 1536 hours.

Blood samples for biochemistry and hematology tests: Screening, day 64 and day 90 post dose.13 Ambulatory blood samples will be collected at 72, 96, 120, 144, 168, 192, 360, 528, 696, 864, 1032, 1200 and 1536 hours post-dose will be collected through fresh vein puncture.

ANOVA will be performed on log transformed Cmax, AUC0-t and AUC0-inf by using SAS or other statistical software.

The following standards for bioequivalence will be applied: The 90% confidence interval of the relative mean Cmax, AUC0-t and AUC0-inf of the test and reference product of Adalimumab should be between 80% and 125% for log-transformed data.

Bearing in mind the complexity of performing a PK profile in subjects in phase I, it is not realistic to establish pre-defined rules for bioequivalence on the basis of the limited blood sampling opportunities and number of subjects in each treatment group.

Pharmacokinetic (PK) Parameters: For Cmax and AUC0-t the 90% confidence interval for the ratio of the test and reference products should be contained within the acceptance interval of 80.00-125.00%.

• Safety assessment: Evaluation and comparison between references vs. test drug in terms of safety end point.

Post study assessment will be done. Physical examination including vital examination, well being assessment, biochemistry and hematology will be done at 64 days and 90 days post dose or on discontinuation of subject from the study.

Part B Part B will be conducted to assess efficacy, tolerability and safety of biosimilar adalimumab (Advixa, Incepta) in compared with reference adalimumab (Humira, AbbVie) in patients with moderate to severe rheumatoid arthritis (RA). Total 160 adult human subjects with moderate to severe active rheumatoid arthritis will be enrolled. 40 mg of either test adalimumab (Advixa) or reference adalimumab (Humira) by subcutaneous route in every two weeks.

The duration of the study will be 12 weeks. A total of eight visits (8) will be scheduled during this study including: screening visit (Visit 0); following screening enrolment Visit 1 (Day 1); Visit 2, Day 15 ± 1; Visit 3, Day 28 ± 3; Visit 4, Day 42 ± 3; Visit 5, Day 56 ± 3; Visit 6, Day 70 ± 3 and Visit 7, Day 84 ± 3.

After each dosage administration, Active/solicited safety follow-up for Adverse Events (either home visit or telephone call 2 times) will be performed for 2 days and passive/un-solicited safety follow-up (spontaneous AE reporting by subject) will be performed for remaining 11 days. This will be repeated after each dosage up to completion of study.

Subjects will be screened for the inclusion/exclusion criteria based on: Demographic data, BMI, clinical history, physical examination (including vital signs), Quantiferon TB gold plus, BNP, ECG, CBC, Chest X-ray (P/A view) (if required based on any significant past medical history and/or positive finding in respiratory system examination), CRP (C- reactive protein), Random blood sugar, Serum bilirubin Total/Direct/Indirect, BUN, Serum urea, ALT (SGPT) blood, AST (SGOT) blood, Alkaline phosphatase serum, Serum creatinine, Serology (hepatitis B, hepatitis C), Urinalysis will be done during the screening.

For female volunteers: In addition to the above tests, urine pregnancy test will be done at the time of screening.

Any other test(s) if required will be done as per the suggestion given by the principal investigator or co-investigator. Blood sample will be collected- For Screening: Before enrollment. For CRP and ESR tests: Day 1, 28, 56 and day 84. For CBC, SGPT, S. Creatinine: Day 28, 56 and day 84 For study completion: Day 84 post dose. Physical examination including vital examination, well-being assessment, Bio-chemistry and hematology tests will be done at day 84 post dose or on discontinuation of subject from the study. For safety evaluation, physical examination and vital examination (Blood pressure, pulse rate, oral temperature and respiratory rate) and Well-being assessment will be done at Screening, day 01, 15 ± 1, 28 ± 3, 42 ± 3, 56 ± 3, 70 ± 3 and day 84 ± 3 post-dose of scheduled time. Bio-chemistry and hematology tests will be reviewed to assess safety of the test drug.

ELIGIBILITY:
Inclusion Criteria:

1. Eligibility of ages for Study: ≥ 18 Years to ≤ 45 Years
2. Genders Eligible for Study: Both
3. Subjects who are able and willing to give written informed consent
4. Willing and able to comply with the requirements of the protocol and be available for the planned duration of the study.

d. Have Chest X ray with no evidence of current active TB or previous (inactive) TB, general infections, heart failure, malignancy, or other clinically significant abnormalities taken at Screening or prior to study and read by a qualified radiologist.

e. Female patients of childbearing potential have to have a negative pregnancy test at the time of screening and agreed to use adequate contraception throughout the study period.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic (Multiple sclerosis), autoimmune, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. Previous history of cancer, except for adequately treated basal cell or squamous cell carcinoma of the skin.
3. Active or latent Tuberculosis or who have a history of Tuberculosis
4. History of invasive systemic fungal infections or other opportunistic infections
5. Systemic or local infection, a known risk for developing sepsis and/or known active inflammatory process
6. Serious infection associated with hospitalization and/or which required intravenous antibiotics
7. History of and/or current cardiac disease or moderate to severe heart failure (NYHA class III/IV).
8. Have received live vaccine(s) within 4 weeks prior to Screening or who will require live vaccine(s) between Screening and the final study visit
9. Intake medication with a half-life > 24 h within 4 weeks or 5 half-lives of the medication prior to investigational product administration
10. Hypersensitivity to the active substance or to any of the excipients (Mannitol and Polysorbate 80)
11. History of severe allergic or anaphylactic reactions to latex
12. History of alcohol, drug, or chemical abuse within 6 months prior to screening
13. History of chronic daily use of narcotic analgesics.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Peak Plasma Concentration (Cmax) of 40 participants will be measured and reported | 6 months
  For "Peak Plasma Concentration (Cmax)", the 90% confidence interval for the ratio of the test and reference products should be contained within the acceptance interval of 80.00-125.00%. and evaluation and comparison between references vs. test drug in terms of safety end point.
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) of 40 participants will be measured and reported | 6 months
  For "Area under the plasma concentration versus time curve (AUC)" , the 90% confidence interval for the ratio of the test and reference products should be contained within the acceptance interval of 80.00-125.00%. and evaluation and comparison between references vs. test drug in terms of safety end point.
For efficacy assessment of 160 patients of Rheumatoid Arthritis, ACR 20 response will be measured and reported in outcome measures result data table | 6 months
  Proportion of patients with an ACR20 response in both the treatment groups at week 12 as well as safety between references vs. test drug should be observed.

CONTACTS AND LOCATIONS:
Overall Officials: Zannat Kawser, M.Phil., Principal Investigator — institute for developing Science and Health initiatives
Locations (1):
- ideSHi, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Schouwenburg PA, van de Stadt LA, de Jong RN, van Buren EE, Kruithof S, de Groot E, Hart M, van Ham SM, Rispens T, Aarden L, Wolbink GJ, Wouters D. Adalimumab elicits a restricted anti-idiotypic antibody response in autoimmune patients resulting in functional neutralisation. Ann Rheum Dis. 2013 Jan;72(1):104-9. doi: 10.1136/annrheumdis-2012-201445. Epub 2012 Jul 3. PMID 22759910
- [Background] Jani RH, Gupta R, Bhatia G, Rathi G, Ashok Kumar P, Sharma R, Kumar U, Gauri LA, Jadhav P, Bartakke G, Haridas V, Jain D, Mendiratta SK. A prospective, randomized, double-blind, multicentre, parallel-group, active controlled study to compare efficacy and safety of biosimilar adalimumab (Exemptia; ZRC-3197) and adalimumab (Humira) in patients with rheumatoid arthritis. Int J Rheum Dis. 2016 Nov;19(11):1157-1168. doi: 10.1111/1756-185X.12711. Epub 2015 Jul 14. PMID 26176644
- [Background] Jamshidi A, Gharibdoost F, Vojdanian M, Soroosh SG, Soroush M, Ahmadzadeh A, Nazarinia MA, Mousavi M, Karimzadeh H, Shakibi MR, Rezaieyazdi Z, Sahebari M, Hajiabbasi A, Ebrahimi AA, Mahjourian N, Rashti AM. A phase III, randomized, two-armed, double-blind, parallel, active controlled, and non-inferiority clinical trial to compare efficacy and safety of biosimilar adalimumab (CinnoRA(R)) to the reference product (Humira(R)) in patients with active rheumatoid arthritis. Arthritis Res Ther. 2017 Jul 20;19(1):168. doi: 10.1186/s13075-017-1371-4. PMID 28728599